CLINICAL TRIAL: NCT05993689
Title: Building TrUst and UNiting Teams Through DouLa partnErship - BUNDLE
Acronym: BUNDLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00047801
Record Dates: First submitted 2023-06-18; First posted 2023-08-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BUNDLE Intervention (Experimental): Proposed components of the intervention will include: 1) attendance at two visits in the 2nd trimester and two visits in the 3rd trimester by a doula; 2) exchange of contact information between the clinic and the doula; 3) exchange of social needs and social-structural risk factors complicating patient's prenatal care from doula and exchange of clinical risk factors complicating prenatal care from obstetric provider; 4) communication between the doula and provider; 5) educating the obstetric team on benefits of doula support; 6) preparing labor and delivery team for presence of doula during labor ; and 7) enhancing doula support postpartum for cardiovascular risk reduction.
  Interventions: Other: BUNDLE
- Usual Care (Active Comparator): Standard of care for pregnancy and pregnancy-related issues will be provided by the obstetric provider as per routine.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: BUNDLE — An integrated model of community-based doulas and clinical obstetric providers
  Arms: BUNDLE Intervention
Other: Usual Care — Standard of care for pregnancy and pregnancy-related issues by the obstetric provider
  Arms: Usual Care

SUMMARY:
The BUNDLE study is a prospective mixed-methods study focused on the early integration of community doula into prenatal care. The study will have three phases: Phase 1 is the qualitative phase of conducting focus groups with Black/African American (AA) birthing people and with medical and community healthcare providers to elicit feedback on how best to integrate community-based doulas and obstetricians into one united model of prenatal care to promote trust and improved maternal health outcomes. Phase 2 tests the effectiveness of the newly developed model on healthcare engagement, trust, and adverse maternal outcomes using randomized control trial of 412 Black/AA pregnant participants. Phase 3 is dissemination of BUNDLE findings in scholarly and community-based forums, including with healthcare leaders and policy makers in Wisconsin, advocating for doula coverage and health system sustainability of the integrated model.

DETAILED DESCRIPTION:
The BUNDLE study is a prospective mixed-methods study focused on the early integration of community doula into prenatal care. The investigators will pursue the following aims using a multidisciplinary team of experts in health disparities, community engagement, qualitative research, maternal-fetal medicine, and doula support:

Aim 1: Develop an integrated prenatal care model of medical providers and community doulas in Southeastern Wisconsin Approach: The investigators will conduct six focus groups with 30 Black/AA birthing people (currently pregnant or recently postpartum) and 30 prenatal healthcare providers (obstetricians, midwives, doulas, social workers, prenatal care coordinators, nurses, mental health providers, and obstetric unit leaders) to elicit feedback on models of doula/medical provider integration with the overarching aim of building trust and improving maternal health outcomes. Focus group findings will be reviewed with a community advisory panel (CAP) developed as part of the Community Partnership of the MCW U54 center, to gain the CAP's input on intervention development.

Aim 2: Compare the effectiveness of the integrated prenatal care model to standard prenatal care in improving healthcare engagement and trust and reducing adverse maternal outcomes Approach: In a two-arm randomized controlled trial conducted at Froedtert and MCW, the investigators will randomize 412 Black/AA pregnant people to BUNDLE or standard prenatal care. Primary outcome is healthcare engagement (starting prenatal care in 1st trimester, attending at least 70% of the recommended visits, attending the postpartum visit, and receipt of recommended vaccination during pregnancy). Secondary outcomes include medical mistrust measured by trust in provider scale, perceived discrimination, and frequencies of severe maternal morbidity as defined by the Centers for Disease Control.

Aim 3: Disseminate findings to scholarly and community-based forums and actively pursue opportunities for systems- and policy-level change Approach: The investigators will disseminate findings regularly in scholarly (conference, grand rounds) and community-based (listening session, town hall) forums. The investigators will leverage the existing partnerships with policymakers, healthcare organizations, and community leaders to implement strategies to sustain successful program outcomes through policy changes at the system and statewide level by advocating for doula coverage and healthcare system sustainability of the integrated prenatal care model.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Black or African American
* Pregnant with singleton gestation
* Has an established OBGY at Froedtert & the Medical College of Wisconsin (F&MCW) Health System

Exclusion Criteria:

* Planning to deliver outside of F&MCW Health System
* Receiving support beyond routing prenatal care, such as group prenatal care or has their own doula
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Healthcare Engagement | From study enrollment and until 12 months postpartum
  A composite of the following variables to assess perinatal healthcare engagement: 1) Attended at least ~75% of the recommended prenatal visits; 2) Attended postpartum visit; 3) Received recommended vaccination during pregnancy.

SECONDARY OUTCOMES:
Trust in Provider | Baseline; third trimester, and postpartum
  A validated 11-item instrument used to measure patients' trust in the provider regarding dependability, confidence, and confidentiality of information.
Reported Discrimination | Baseline, third trimester and postpartum
  Measured with a validated survey of patient self-report on how often in the past 12 months, individuals felt treated poorly due to race.
Perceived Stress | Baseline, third trimester and postpartum
  Measured with Cohen's Perceived Stress Scale
Depression | Baseline, third trimester and postpartum
  Measured with the Patient Health Questionnaire-9 (PHQ-9)
Cesarean birth | At study completion
  Cesarean birth for any indication other than prior cesarean
Unplanned healthcare utilization | Up to 12 months postpartum
  Prenatal or postpartum (up to 12 weeks postpartum) unplanned emergency room visits or hospitalizations.
Severe Maternal Morbidity | Up to 12 months postpartum
  Composite outcome of the following diagnoses using ICD-10 codes: acute myocardial infarction, aneurysm, acute renal failure, adult respiratory distress syndrome, amniotic fluid embolism, cardiac arrest, disseminated intravascular coagulation, eclampsia, heart failure, puerperal cerebrovascular disorders, pulmonary edema, severe anesthesia complications, sepsis, shock, sickle cell disease with crisis, air and thrombotic embolism blood products transfusion, hysterectomy, temporary tracheostomy, ventilation.
Breastfeeding Initiation | Up to 12 months postpartum
  Rates of breastfeeding initiation prior to discharge from the hospital
Group-Based Medical Mistrust Scale | Baseline; Week 27 up to birth (third trimester); Birth up to Week 40 (Postpartum)
  A 12-item validated survey focused on healthcare provided in the social context of racism and discrimination.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States